CLINICAL TRIAL: NCT02636244
Title: A Multi-Center, Open-Label Phase 2 Study to Evaluate the Safety and Efficacy of SHAPE Gel, a Histone Deacetylase Inhibitor, in Patients With Alopecia Areata
Brief Title: Safety and Efficacy Study of SHAPE Gel in Alopecia Areata
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP-141-POC-0004-PTL
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHAPE Gel (Experimental): 1% SHAPE Gel applied twice daily for 12 weeks.
  Interventions: Drug: SHAPE Gel

INTERVENTIONS:
Drug: SHAPE Gel
  Other Names: SHP-141

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SHAPE Gel applied topically to adult patients with alopecia areata of the scalp.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of scalp alopecia areata and scalp hair loss due to alopecia areata for a minimum of six months and a maximum of two years.
* Patients taking thyroid medication or hormonal therapy must be on a stable dose for 6 months and maintain such throughout the study.
* Willingness to maintain same hair style, including shampoo and hair dye, throughout the study period.
* Willingness to have a small micro dot tattoo placed to allow for photographic analysis of treatment and application of study medication.

Exclusion Criteria:

* History of systemic or cutaneous malignancy and/or lymphoproliferative disease, other than patients with: up to 3 basal cell carcinoma; up to three well differentiated cutaneous squamous cell carcinoma; and/or cervical intraepithelial neoplasm (CIN), treated successfully with no evidence of disease, and treated for greater than 6 months prior to study entry.
* Current actinic keratosis on the scalp and/or face
* Nevi or cutaneous lesions thought suspicious for malignancy.
* History of or current gastrointestinal, pulmonary, cardiovascular, genitourinary or hematological disease, CNS disorders, infectious disease or coagulation disorders that would preclude participation in and completion of study assessments.
* Positive for hepatitis B surface antigen, HIV or hepatitis C.
* Co-existent androgenetic alopecia: in males: Norwood-Hamilton stage IV, V or VI; in females: Ludwig stage II or III.
* Unwillingness to discontinue use of non-breathable wigs, weaves or shaving of scalp throughout course of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-08 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Response evaluated using modified Severity of Alopecia Tool (mSALT) | Every 4 weeks; up to 24 weeks
  Severity of Alopecia Tool (SALT) estimates percent scalp hair loss and percent regrowth of hair following intervention

SECONDARY OUTCOMES:
Effects on quality of life using Subject Assessment of Hair Loss (SAHL) | Every 4 weeks; up to 24 weeks
  The SAHL compares baseline hair volume and hair density with end of treatment hair volume and density
Effects on quality of life using Alopecia Areata Symptom Impact Scale (AASIS) | Every 4 weeks; up to 24 weeks
  AASIS rates the severity of alopecia areata symptoms and interference of alopecia areata with daily functioning
Effects on quality of life using the Skindex-16 | Every 4 weeks; up to 24 weeks
  Skindex-16 assesses how often symptoms or signs of alopecia areata have been bothersome
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | Every 4 weeks, up to 12 weeks
  Evaluation of safety and tolerability will be assessed through adverse events (AEs), vital signs, physical examination, assessment of local skin changes and changes in clinical laboratory parameters

OTHER OUTCOMES:
Pharmacodynamic effect determined through assessment of lymphocyte subsets | Up to 12 weeks
  Measured by CD3, CD4 and CD8 lymphocytes in skin as well as by other assessments of immune modulation in the scalp